CLINICAL TRIAL: NCT02654743
Title: An Examination of Changes in Urinary Metabolites With Use of an Antioxidant Supplement, Sulforaphane, in School-aged Children With Autism
Brief Title: Open Label of Clinical Trial of Sulforaphane in Children With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF15-17002
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SF (Experimental): Sulforaphane (SF) will be administered in an approximate dosage of 1 µmol SF/lb (2.2 kg µmol/kg) body weight. This dosage roughly approximates the dosage that was used in the Singh et al, (2014; PNAS) clinical trial of sulforaphane in male adolescents and adults with autism. The sulforaphane will be supplied as glucoraphanin (GR)-enriched broccoli seed extract tablets (manufacturing details follow). Each active tablet will contain 125 mg broccoli seed extract (containing 37 µmol GR, which is equivalent to about 15 µmol SF), 50 mg dried broccoli sprouts (a source of myrosinase, the enzyme that converts GR to SF), 15 mg ascorbic acid, 55.90 mg microcrystalline cellulose, and other minor GRAS excipients used for tablet forming.
  The total dose per day will depend of study participants' body weight.
  Interventions: Dietary Supplement: Sulforaphane

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Children with ASD will receive Sulforaphane in this study

SUMMARY:
This is an open-label, 4-month study examining the effects of Sulforaphane (SF) on behavior in children with ASD and the correlation between behavior change and urinary metabolites. The goal is to determine a potential mechanism of action of SF in this population.

DETAILED DESCRIPTION:
Sulforaphane (SF) is an isothiocyanate found in high levels in crucifers belonging to the family Brassicaceae (including broccoli, cabbage, cauliflower, brussels sprouts, Chinese cabbage and turnips). Many previous studies have documented that consumption of these vegetables is associated with a reduced risk of cancer (lung, breast, colon, rectum, and prostate).(Juge et al. 2007) The mechanism of action of these beneficial effects is believed to be due to the ability of SF to up-regulate genes that improve cellular response to oxidative stress, inflammation, DNA-damaging electrophiles, and radiation.(Singh et al. 2014) In a recent small, randomized controlled trial in children with autism, SF was shown to have beneficial effects on aberrant and social behavior.(Singh et al. 2014) The mechanism of action of this beneficial effect has not been established in children with ASD. Our primary goal is to examine changes in urinary metabolites in children with autism who receive SF to determine if changes in behavior are associated with changes in urinary metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, enrolled at OHS, age 6-22 and with a diagnosis of ASD.
* ASD diagnosis will be established by standard criteria (DSM-IV criteria and expert clinician review of medical records and child observation).
* Written informed consent obtained from the subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Urinary metabolites | 3 month
  Urine samples will be analyzed by lab and result will be provided
Behavior Measures | 3 months
  Measuring behavior using ABC (Aberrant Behavior Checklist)- self reported 58 questions from 0-3 scale (0-not a problem; 3=severe problem)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hendren, DO, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bent S, Lawton B, Warren T, Widjaja F, Dang K, Fahey JW, Cornblatt B, Kinchen JM, Delucchi K, Hendren RL. Identification of urinary metabolites that correlate with clinical improvements in children with autism treated with sulforaphane from broccoli. Mol Autism. 2018 May 30;9:35. doi: 10.1186/s13229-018-0218-4. eCollection 2018. PMID 29854372